CLINICAL TRIAL: NCT02068651
Title: A Community-based Advance Care Planning Programme to Improve End-of-life Care in Patients With Advanced Disease: A Mixed-method Approach
Brief Title: A Community-based Advance Care Planning Programme for Patients With Advanced Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Food and Health Bureau, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Dr. Helen YL Chan, Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 11120861
Record Dates: First submitted 2014-02-13; First posted 2014-02-21 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Disease
Keywords: End-of-life care; Treatment decision making; Advance care planning
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Advance care planning programme (Experimental): Participants in the experimental group will receive a structured advance care planning programme, namely Let Me Talk, delivered by a trained nurse facilitator. The programme will be conducted on individual basis through three one-hour home visits, once weekly. Family carers of the participants will be invited to all sessions.
  Interventions: Behavioral: Advance care planning programme
- Usual care (No Intervention): Participants in the control group will receive three weekly home visits with basic health assessment and education provided by the trained nurse facilitator. If they request advance care planning information or assistance, an advance directive form, which is available on the Internet for public access, will be provided to them for their information.

INTERVENTIONS:
Behavioral: Advance care planning programme — It is a multi-faceted programme which includes an educational component with support of multimedia materials, reflection on personal values and a facilitated discussion between patient and family carer over future care. It will be delivered to each pair of participant and family carer on individual basis. By the end of the programme, each participant will have a personal workbook summarising the advance care planning process for record.
  Arms: Advance care planning programme

SUMMARY:
Advance care planning has been recommended as an integral part of care for patients with life-limiting disease, but relevant development in Hong Kong is still in its infancy. This proposed study attempts to address this service gap by promoting advance care planning to patients with advanced disease. It is hypothesized that the proportion of patients whose end-of-life care preferences were known in the experimental group will be significantly higher than that in the control group.

DETAILED DESCRIPTION:
This study aims to evaluate the impacts of a community-based advance care planning programme on end-of-life care of patients with advanced disease. A mixed-method approach, including a randomized controlled trial and qualitative interviews, will be used. Participants in the experimental group will received a structured advance care planning programme delivered by a trained facilitator. It includes an educational component, reflection and a family meeting.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above
* meet one of the three triggers for supportive /palliative care as suggested in the Gold Standards Framework
* living at home
* being communicable

Exclusion Criteria:

* mentally incompetent
* cannot nominate a family carer
* have already signed an advance directive
* have been referred to palliative care service

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2014-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
End-of-life care preferences | 6 months
  In this study, end-of-life care preferences include goal for end-of-life care and decisions over the use of life-sustaining treatments relevant to individual's anticipated health changes. So, whether the patients' end-of-life care preferences is known at different timepoints will be determined based on (1) the congruence between patients' end-of-life care preferences and family carers' predicted end-of-life care preferences for patients; and (2) whether patients' end-of-life preferences are documented in their medical record.

SECONDARY OUTCOMES:
Level of certainty about future care | 6 months
  The SURE test (Legare, Kearing, Clay, Gagnon, D'Amours, Rousseau & O'Connor, 2010) will be used to measure the patient's level of decisional conflict in making decisions related to future care. Patients will be asked to rate their certainty in their future care on four items by using a dichotomous response format: yes or no. Good construct validity and reliability were demonstrated. It has previously been translated into Chinese and tested among local older people .
Health care utilization | 6 months
  Patient's medical records will be retrieved retrospectively six months after their enrolment to review their health care utilization over the study period, including the number of visits to the emergency department, unplanned admission, length of hospital stay, as well as investigation, procedures and treatment received.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Chan, RN PhD, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong; Diana Lee, RN PhD, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong; Carmen Chan, RN PhD, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong; Iris Lee, RN PhD, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong; Doris Leung, PhD, Principal Investigator — The Nethersole School of Nursing, The Chinese University of Hong Kong
Locations (1):
- Haven of Hope Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No